CLINICAL TRIAL: NCT03787654
Title: Effect of Electroacupuncture for Women With Urgency-predominant Mixed Urinary Incontinence: a Three Armed Non-inferior Randomized Controlled Trial
Brief Title: Electroacupuncture and Solifenacin for Urgency-predominant Mixed Urinary Incontinence
Acronym: EASE-UMUI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Principle investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-163-KY
Record Dates: First submitted 2018-12-22; First posted 2018-12-26 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Mixed Urinary Incontinence; Urgency-predominant Mixed Urinary Incontinence
MeSH Terms: interventions — Electroacupuncture; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: participants in electroacupuncture and sham electroacupuncture groups are blinded, and solifenacin group is open.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- electroacupuncture group (Experimental): Acupoints of bilateral Zhongliao (BL33), Huiyang (BL35) and Sanyinjiao (SP6) are stimulated by Huatuo Brand disposable needles and SDZ-V electronic apparatus.
  Interventions: Device: electroacupuncture
- sham electroacupuncture group (Sham Comparator): Sham acupoints 1 cun(≈15mm) horizontally outwardly lateral to BL33 and BL35, and 0.5 cun(≈10mm) horizontally behind SP6 are stimulated superficially with a small electricity current by needles of 0.30×40mm size and SDZ-V electronic apparatus.
  Interventions: Device: sham electroacupuncture
- Solifenacin group (Active Comparator): subjects will orally take Solifenacin 5-10mg per day.
  Interventions: Drug: Solifenacin

INTERVENTIONS:
Device: electroacupuncture — BL33 and BL35 are inserted by needles of 0.30×75mm size till a depth of 60~70mm. SP6 is inserted by needle of 0.30×40mm size till a depth of 25-30mm. After manipulation and deqi sensation generation, the electrodes will be attached to the acupoints transversely with 20Hz continuous wave and an electricity current of 2mA-6.5mA at BL33 and BL35, and 1-3.5mA at SP6. The current is adjusted from zero to the degree where patients can tolerate.
  Subjects receive 3 sessions per week（every other day ideally) for 12 weeks, 36 sessions in total.
  Other Names: EA group
  Arms: electroacupuncture group
Device: sham electroacupuncture — In sham electroacupuncture group, sham acupoints 1 cun(≈15mm） horizontally outwardly lateral to BL33 and BL35, and 0.5 cun (≈10mm) horizontally behind SP6 are stimulated by needles of 0.30×40mm size. The needles are inserted to a depth of 2-3mm to stand still, without any manipulation and sensation of deqi. The electrodes will also be attached to needles with an electricity current of 0.1-0.3mA.
  The sessions will be the same as the electroacupuncture group.
  Other Names: SEA group
  Arms: sham electroacupuncture group
Drug: Solifenacin — Subjects take solifenacin 5-10mg per day for a succession of 36 weeks. The dose change is decided by doctors under a comprehensive consideration of side effects and Patient Global Symptom Control (PGSC), which is applied to evaluate the effectiveness of Solifenacin at the 4th, 8th, 12th and 24th week.The medicine can be discontinued at any time if the adverse effect is rather severe.
  Other Names: Drug group
  Arms: Solifenacin group

SUMMARY:
The study is to determine the effect of electroacupuncture in female patients with urgency-predominant mixed urinary incontinence. A three-arm non-inferior randomized controlled trial (RCT) using electroacupuncture, sham electroacupuncture and solifenacin with a total sample of 282 is proposed.

The hypothesis is that the improvement (difference in number of urgency urinary incontinence episodes between baseline and 12-week evaluation) in the electroacupuncture group would be 50% or less of the difference in the improvement between the Solifenacin and the sham electroacupuncture groups.

DETAILED DESCRIPTION:
Mixed urinary incontinence (MUI) features complaint or involuntary loss of urine associated with urgency and also with effort or physical exertion or on sneezing or coughing. It is regarded as urgency-predominant mixed urinary incontinence (UMUI) when sudden sensation of voiding accompanied by uncontrolled incontinence domains the symptoms. UMUI can bring shame and inconvenience to patients.

As first-line medicine for urge-predominant urinary incontinence, Solifenacin can reduce urgency urinary incontinence episodes in 24 hours. However, the side effects tend to bring about poor compliance among patients.

Acupuncture might be effective in treating UMUI. Previous research indicated that electroacupuncture might be noninferior to pelvic floor muscle training plus Solifenacin in reducing the urgency incontinence episodes of UMUI women. However, that study didn't focuse on UMUI exclusively, thus unable to decide whether electroacupuncture is effective in the treatment of UMUI.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients diagnosed with mixed urinary incontinence in accordance with EAU guideline by history intaking and physical examination[8];
2. Age between 18 and 80 years old;
3. Urgency index greater than stress index by MESA questionnaire[12];
4. At least 4 episodes of urgency urinary incontinence in 72-hour voiding diary;
5. With MUI for at least 3 months, and more than 50% of the total incontinence episodes is urgency one in 72-hour voiding diary;
6. Positive cough test;
7. A voluntarily-signed written informed content.

Exclusion Criteria:

1. Having pure stress urinary incontinence, pure urgency urinary incontinence, overflow urinary incontinence or neurogenic bladder;
2. Uncontrolled urinary tract infection;
3. Tumor in urinary system or pelvic organs;
4. Pelvic organ prolapse≥degreeⅡ;
5. Residual urine volume≥100ml;
6. Maximum flow rate<15ml/s;
7. Treated incontinence by acupuncture or positive medications, such as antimuscarinic drug within the past 1 month;
8. Underwent surgery of anti-incontinence or in pelvic area, metrectomy included;
9. Complication of uncontrolled diabetes and severe hypertension;
10. Complicated diseases in nerves system that could hamper hypourethral function, such as Multiple sclerosis, senile dementia, Parkinson's disease, spinal cord injury, cauda equina nerve injury and multiple system atrophy;
11. Severe complications in cardiac, lungs, cerebrum, hepar, renal system, psychonosology and coagulation function, or obvious cognitive disability;
12. Installed a cardiac pacemaker;
13. Allergic to solifenacin or with contraindications to antimuscarinic drug, like urinary retention, gastrointestinal peristalsis paralysis, myasthenia gravis, ulcerative colitis, angle-closure glaucoma;
14. Allergic to metal or intolerant to the stimulation of electroacupuncture;
15. Already with child or plan to conceive in the future 1 year, or within 1 year after delivery.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of urgency urinary incontinence episodes in average 24 hours from baseline based on 3-day voiding diary. | week 12
  3-day voiding diary is a reliable objective method to quantify the incontinence episode frequency and are a sensitive measurement to monitor the treatment response. In voiding diary, voiding episodes, urgency episodes, incontinence episodes, the volume drunk and the pads consumed are all recorded.

SECONDARY OUTCOMES:
Change of urgency urinary incontinence episodes in average 24 hours from baseline based on 3-day voiding diary. | week 4, week 8, week 24, week 36
  3-day voiding diary is a reliable objective method to quantify the incontinence episode frequency and are a sensitive measurement to monitor the treatment response. In voiding diary, voiding episodes, urgency episodes, incontinence episodes, the volume drunk and the pads consumed are all recorded.
Change of urinary incontinence episodes in average 24 hours from baseline based on 3-day voiding diary. | week 4, week 8, week 12, week 24, week 36
  3-day voiding diary is a reliable objective method to quantify the incontinence episode frequency and are a sensitive measurement to monitor the treatment response. In voiding diary, voiding episodes, urgency episodes, incontinence episodes, the volume drunk and the pads consumed are all recorded.
Proportion of subjects with at least 50% reduce of urgency urinary incontinence episodes in average 24 hours compared with baseline based on 3-day voiding diary. | week 4, week 8, week 12, week 24, week 36
  3-day voiding diary is a reliable objective method to quantify the incontinence episode frequency and are a sensitive measurement to monitor the treatment response. In voiding diary, voiding episodes, urgency episodes, incontinence episodes, the volume drunk and the pads consumed are all recorded.
Proportion of subjects with complete resolution of urgency urinary incontinence episodes in average 24 hours based on 3-day voiding diary. | week 4, week 8, week 12, week 24, week 36
  3-day voiding diary is a reliable objective method to quantify the incontinence episode frequency and are a sensitive measurement to monitor the treatment response. In voiding diary, voiding episodes, urgency episodes, incontinence episodes, the volume drunk and the pads consumed are all recorded.
Proportion of subjects with at least 50% reduce of urinary incontinence episodes in average 24 hours compared with baseline based on 3-day voiding diary. | week 4, week 8, week 12, week 24, week 36
  3-day voiding diary is a reliable objective method to quantify the incontinence episode frequency and are a sensitive measurement to monitor the treatment response. In voiding diary, voiding episodes, urgency episodes, incontinence episodes, the volume drunk and the pads consumed are all recorded.
Change of voiding episodes in average 24 hours from baseline based on 3-day voiding diary. | week 4, week 8, week 12, week 24, week 36
  3-day voiding diary is a reliable objective method to quantify the incontinence episode frequency and are a sensitive measurement to monitor the treatment response. In voiding diary, voiding episodes, urgency episodes, incontinence episodes, the volume drunk and the pads consumed are all recorded.
Change of voiding episodes graded as 3/4 in average 24 hours from baseline based on the Patient Perception of Intensity of Urgency Scale( PPIUS). | week 4, week 8, week 12, week 24, week 36
  Patient Perception of Intensity of Urgency Scale (PPIUS) is recommended by the European Medicines Agency to grade the urgency of voiding. Voiding graded at 1 and 2 levels of urgency are regarded as normal or strong desire to void rather than urgency, while 3 and 4 levels are regarded as urgency episodes.
Change of nocturia episodes in average 24 hours from baseline based on 3-day voiding diary. | week 4, week 8, week 12, week 24, week 36
  3-day voiding diary is a reliable objective method to quantify the incontinence episode frequency and are a sensitive measurement to monitor the treatment response. In voiding diary, voiding episodes, urgency episodes, incontinence episodes, the volume drunk and the pads consumed are all recorded.
Change of pad consuming in average 24 hours from baseline based on 3-day voiding diary. | week 4, week 8, week 12, week 24, week 36
  3-day voiding diary is a reliable objective method to quantify the incontinence episode frequency and are a sensitive measurement to monitor the treatment response. In voiding diary, voiding episodes, urgency episodes, incontinence episodes, the volume drunk and the pads consumed are all recorded.
volume change of water intake in average 24 hours from baseline based on 3-day voiding diary. | week 4, week 8, week 12, week 24, week 36
  3-day voiding diary is a reliable objective method to quantify the incontinence episode frequency and are a sensitive measurement to monitor the treatment response. In voiding diary, voiding episodes, urgency episodes, incontinence episodes, the volume drunk and the pads consumed are all recorded.
Change of International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI-SF ) score from baseline. | week 4, week 8, week 12, week 24, week 36
  ICIQ-UI-SF was a questionnaire developed by the International Consultation on Incontinence to evaluate the severity of incontinence and impact to QoL in the past four weeks. It contains four items: frequency, amount of leakage, impact of UI on QoL and a separate item to indicate the cause of incontinence. The score was the sum of the first three items, providing a total score ranging from 0 to 21 with a higher score indicating worse symptoms and greater impact on QoL.
Change of Overactive bladder questionnaire short form (OABq-SF) score from baseline. | week 4, week 8, week 12, week 24, week 36
  OABq-SF is a validated questionnaire to assess the bother of OAB symptoms and effect on QoL in the past four weeks. It includes coping, sleep and emotional interaction. The scores were transformed to a 0- to 100-point scale, and higher scores on the symptom-severity scale indicate worse symptoms, whereas higher scores on the QoL scale indicate better quality of life.
Proportion of subjects with adequate improvement assessed by Patient global impression improvement (PGI-I). | week 12, week 36
  Patient global impression improvement (PGI-I) is a scale range from 1 to 7, with 1 indicating very much better and 7 indicating very much worse. Adequate improvement is defined as a rating of 1 or 2 by PGI-I.
Change of residual urinary volume from baseline tested by abdominal B-ultrasound. | week 12
  Abdominal B-ultrasound is objective way to test the residual urinary volume.

OTHER OUTCOMES:
Proportion of subjects bearing expectancy towards acupuncture AND proportion of subjects bearing expectancy towards drugs. | baseline
  Expectancy of acupuncture and drugs will be recorded at baseline. Participants in the electroacupuncture and sham electroacupuncture groups will be asked to answer: "Do you think acupuncture is effective in improving the symptoms of incontinence?" Subjects will choose answer from "Have no idea", "Yes" or "No".
  Participants in the solifenacin group will be asked to answer: "Do you think drug is effective in improving the symptoms of incontinence?" Subjects will choose answer from "Have no idea", "Yes" or "No".
Proportion of subjects successfully blinded | week 12
  Within 5 minutes after any treatment in week 12, subjects will be asked the question that: "Do you think you have received traditional electroacupuncture in the past 12 weeks?" Answer will be chosen from "Yes" or "No". The answer of "yes" indicates successful blinding.
Incidence of adverse events | week 0-36
  Side effects induced by Solifenacin mainly include dry mouth, dry eye and constipation.
  Unintended events and feelings related to EA and SEA include broken needles, fainting, bleeding, bruising, infection and aposteme, unbearable ache (VAS≥8), vomiting, nausea, palpitations, dizziness, headache, anorexia and insomnia, etc.
  Adverse events irrelevant with the treatment will also be recorded in detail.

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, PhD, Principal Investigator — Guanganmen Hospital
Locations (1):
- Guang An Men Hospital, Beijing, China

REFERENCES:
- [Derived] Sun Y, Liu Y, Su T, Sun J, Wu Y, Liu Z. Electroacupuncture versus solifenacin for women with urgency-predominant mixed urinary incontinence: a protocol for a three-armed non-inferiority randomized controlled trial. BMC Complement Med Ther. 2020 Jan 23;20(1):18. doi: 10.1186/s12906-019-2784-1. PMID 32020889